CLINICAL TRIAL: NCT01417052
Title: A Phase 1, Single-Center, Randomized, Double-Blind, Placebo-Controlled, Dose Escalation Study to Determine the Safety and Efficacy of Daily Orally Administered LX3305 in Subjects With Active Rheumatoid Arthritis (RA)
Brief Title: A Study to Determine the Safety and Efficacy of LX3305 in Subjects With Active Rheumatoid Arthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lexicon Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LX3305.1-106-RA; LX3305.106 (Other: Lexicon Pharmaceuticals, Inc.)
Record Dates: First submitted 2011-08-12; First posted 2011-08-16 (Estimated); Last update posted 2012-08-02 (Estimated); Status verified 2012-08

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (10):
- 50 mg LX3305 QD (Experimental)
  Interventions: Drug: 50 mg LX3305 QD
- 100 mg LX3305 QD (Experimental)
  Interventions: Drug: 100 mg LX3305 QD
- 150 mg LX3305 QD (Experimental)
  Interventions: Drug: 150 mg LX3305 QD
- 200 mg LX3305 QD (Experimental)
  Interventions: Drug: 200 mg LX3305 QD
- 250 mg LX3305 QD (Experimental)
  Interventions: Drug: 250 mg LX3305 QD
- 300 mg LX3305 QD (Experimental)
  Interventions: Drug: 300 mg LX3305 QD
- 400 mg LX3305 QD (Experimental)
  Interventions: Drug: 400 mg LX3305 QD
- 250 mg LX3305 BID (Experimental)
  Interventions: Drug: 250 mg LX3305 BID
- 500 mg LX3305 QD (Experimental)
  Interventions: Drug: 500 mg LX3305 QD
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 50 mg LX3305 QD — 50 mg LX3305 once daily in capsule form
  Arms: 50 mg LX3305 QD
Drug: 100 mg LX3305 QD — 100 mg LX3305 once daily in capsule form
  Arms: 100 mg LX3305 QD
Drug: 150 mg LX3305 QD — 150 mg LX3305 once daily in capsule form
  Arms: 150 mg LX3305 QD
Drug: 200 mg LX3305 QD — 200 mg LX3305 once daily in capsule form
  Arms: 200 mg LX3305 QD
Drug: 250 mg LX3305 QD — 250 mg LX3305 once daily in capsule form
  Arms: 250 mg LX3305 QD
Drug: 300 mg LX3305 QD — 300 mg LX3305 once daily in capsule form
  Arms: 300 mg LX3305 QD
Drug: 400 mg LX3305 QD — 400 mg LX3305 once daily in capsule form
  Arms: 400 mg LX3305 QD
Drug: 250 mg LX3305 BID — 250 mg LX3305 twice daily in capsule form
  Arms: 250 mg LX3305 BID
Drug: 500 mg LX3305 QD — 500 mg LX3305 once daily in capsule form
  Arms: 500 mg LX3305 QD
Drug: Placebo — Matching placebo dosing in capsule form
  Arms: Placebo

SUMMARY:
The primary objective of this study is to determine the safety of LX3305 in a dose escalation compared with placebo over 12 weeks in subjects with active rheumatoid arthritis (RA).

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects, aged 18 to 75 years
* Active rheumatoid arthritis (RA), class I to III (defined by the American College of Rheumatology), diagnosed at least 3 months prior to Screening
* Minimum of 4 swollen joints (at Screening and Day 1), minimum of 4 tender joints (at Screening and Day 1), and serum C-reactive protein (CRP) level >1.2x the upper limit of normal and/or elevated erythrocyte sedimentation rate (ESR)
* If receiving methotrexate (7.5 mg to 25 mg/week), subject must have been treated for at least 6 weeks prior to Screening and currently receiving a stable dose of methotrexate (MTX) with a stable route of administration, and have no plans to change MTX dose during the study
* Ability to give written informed consent

Exclusion Criteria:

* Women who are pregnant or nursing
* RA diagnosis prior to 16 years of age (juvenile RA)
* Intra-articular and/or parenteral corticosteroids within 4 weeks of study Day 1
* Receipt of live vaccine within 4 weeks prior to Day 1
* Major surgical procedure within 8 weeks prior to Day 1
* Blood donation within 4 weeks prior to Day 1
* Any systemic inflammatory condition
* History of bleeding diathesis
* History of medically significant opportunistic infection
* History of drug or alcohol abuse within 3 years prior to Day 1
* History of cancer within 5 years prior to Day 1
* Presence of hepatic or biliary disease
* History of tuberculosis
* History of human immunodeficiency virus (HIV)
* Any clinically significant laboratory test results, in the opinion of the investigator
* Use of any investigational agent or participation in an investigative trial within 30 days of Day 1
* Concurrent use of any biologic agent for the treatment of RA or concomitant disease modifying antirheumatoid drugs (other than MTX, hydroxychloroquine, leflunomide, and sulfasalazine - at stables doses for 8 weeks)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-09; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Number of subjects experiencing an adverse event (AE) | 14 weeks

SECONDARY OUTCOMES:
Change from baseline in absolute lymphocyte counts | 14 weeks
Maximum observed plasma concentration | 14 weeks
Time at which maximum observed plasma concentration occurs | 14 weeks
Half-life of drug in plasma | 14 weeks
Changes from baseline in global health | 14 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Joel Freiman, MD, MPH, Study Director — Lexicon Pharmaceuticals, Inc.
Locations (1):
- Lexicon Investigational Site, Dallas, Texas, United States